CLINICAL TRIAL: NCT02442466
Title: Proof of Concept Study With an Endothelin Receptor B Inhibitor (BQ-788) for Human Melanoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulties to recruit on time the required patient population.
Sponsor: MelCure SA (Industry)
Collaborators: California Institute of Technology (Other); University of Bern (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: MelCure
Record Dates: First submitted 2015-04-26; First posted 2015-05-13 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Endothelin receptor B inhibitor BQ-788 (Experimental): Intra-lesion administration of an Endothelin Receptor B inhibitor (BQ-788)
  Interventions: Drug: Endothelin Receptor B inhibitor BQ788
- PBS (Experimental): Intra-lesion administration of vehicle
  Interventions: Drug: PBS

INTERVENTIONS:
Drug: Endothelin Receptor B inhibitor BQ788
  Arms: Endothelin receptor B inhibitor BQ-788
Drug: PBS
  Arms: PBS

SUMMARY:
Intra-lesion administration of an Endothelin Receptor B inhibitor (BQ-788) or vehicle was preformed in 5 melanoma patients to have a preliminary analysis of safety, dose, duration and relevance of results observed in pre-clinical studies to the human disease.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed consent
* Histologically confirmed melanoma
* Disease stage III or IV
* At least 2 injectable and surgically removable cutaneous metastasis
* Age > 18 years
* Clinically stable medical condition

Exclusion Criteria:

* Primary ocular melanoma
* Symptomatic intracranial melanoma
* History of severe neurological, cardiovascular, renal, hepatic, endocrinological, respiratory, bone marrow, autoimmune or infectious (HIV) disease
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Tumour response by size measurement and histological examination | 3 to14 days

SECONDARY OUTCOMES:
Measuring changes in tumor cell proliferation by histological analyses using Ab staining | 3 to 14 days
Evaluation of changes in mRNA as well as protein expression levels of Endothelin Receptor B by PCR and Ab staining | 3 to 14 days
Evaluation of changes in blood vessels formation by histological examination using Ab staining | 3 to 14 days
Evaluation of changes in immune cell infiltration by histological examination using Ab staining | 3 to 14 days

REFERENCES:
- [Background] Lahav R, Ziller C, Dupin E, Le Douarin NM. Endothelin 3 promotes neural crest cell proliferation and mediates a vast increase in melanocyte number in culture. Proc Natl Acad Sci U S A. 1996 Apr 30;93(9):3892-7. doi: 10.1073/pnas.93.9.3892. PMID 8632985
- [Background] Lahav R, Dupin E, Lecoin L, Glavieux C, Champeval D, Ziller C, Le Douarin NM. Endothelin 3 selectively promotes survival and proliferation of neural crest-derived glial and melanocytic precursors in vitro. Proc Natl Acad Sci U S A. 1998 Nov 24;95(24):14214-9. doi: 10.1073/pnas.95.24.14214. PMID 9826680
- [Background] Lahav R, Heffner G, Patterson PH. An endothelin receptor B antagonist inhibits growth and induces cell death in human melanoma cells in vitro and in vivo. Proc Natl Acad Sci U S A. 1999 Sep 28;96(20):11496-500. doi: 10.1073/pnas.96.20.11496. PMID 10500205
- [Background] Lahav R, Suva ML, Rimoldi D, Patterson PH, Stamenkovic I. Endothelin receptor B inhibition triggers apoptosis and enhances angiogenesis in melanomas. Cancer Res. 2004 Dec 15;64(24):8945-53. doi: 10.1158/0008-5472.CAN-04-1510. PMID 15604257
- [Background] Lahav R. Endothelin receptor B is required for the expansion of melanocyte precursors and malignant melanoma. Int J Dev Biol. 2005;49(2-3):173-80. doi: 10.1387/ijdb.041951rl. PMID 15906230
- [Derived] Wouters J, Hunger RE, Garrod T, Dubuis B, Hunziker T, van den Oord JJ, Lahav-le Coutre R. First-in-Human Proof-of-Concept Study: Intralesional Administration of BQ788, an Endothelin Receptor B Antagonist, to Melanoma Skin Metastases. Oncologist. 2015 Oct;20(10):1121-2. doi: 10.1634/theoncologist.2015-0139. Epub 2015 Sep 1. PMID 26330458